CLINICAL TRIAL: NCT07171190
Title: Targeted Abdominal CT in Conjunction With Lung Cancer Screening - a Pilot Study (TACTICAL1): a Randomised Controlled Pilot Study of Adding Abdominal Non-contrast CT to Lung Cancer Screening CT Thorax Amongst High Lung Cancer Risk Ever-smokers Aged 55-70.
Brief Title: Targeted Abdominal CT in Conjunction With Lung Cancer Screening
Acronym: TACTICAL1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Grant Stewart, Professor Grant Stewart, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: G128732
Record Dates: First submitted 2025-08-14; First posted 2025-09-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer); Kidney Cancers; AAA - Abdominal Aortic Aneurysm; Renal Stones
Keywords: Screening; NHS Lung Cancer Screening; Kidney cancer; Abdominal cancer; Lung cancer; Abdominal Aortic Aneurysms (AAA); Abdominal screening
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Aortic Aneurysm, Abdominal; Nephrolithiasis; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Invitation control arm (Active Comparator): Invited to NHS Lung Cancer Screening to assess lung cancer risk via letter or text message, following the normal process
  Interventions: Other: Lung Cancer Screening Invitation Intervention
- Invitation intervention arm (Experimental): Will have additional text included in the standard Lung Cancer Screening letter or text explaining that, if eligible, they may also be offered a scan of their abdomen at the same time as their lungs.
  Interventions: Other: Lung Cancer Screening Invitation Intervention
- Scan control arm (Active Comparator): For the scan control batches, those who are 'high risk' following the LCS assessment will have an appointment booked for LCS in the normal way by the LCS assessor.
  Interventions: Diagnostic Test: Abdominal scan intervention
- Scan intervention arm (Experimental): Those who are 'high risk' following the LCS assessment will be invited to have an abdominal CT scan at the same time as their lung scan.
  Interventions: Diagnostic Test: Abdominal scan intervention

INTERVENTIONS:
Other: Lung Cancer Screening Invitation Intervention — Participants are invited to the NHS Lung Cancer Screening to assess lung cancer risk via letter or text message
  Arms: Invitation control arm; Invitation intervention arm
Diagnostic Test: Abdominal scan intervention — Receiving an abdominal CT scan at the same time as the lung scan.
  Arms: Scan control arm; Scan intervention arm

SUMMARY:
Early detection through screening can improve cancer survival by identifying it when it's most treatable. The NHS now offers Lung Cancer Screening (LCS) assessments to people aged 55-74 who have ever smoked. Those at higher risk of lung cancer are offered a lung scan.

This group also has a high risk of developing abdominal cancers, such as kidney cancer. A recent study explored whether it would be feasible to extend the lung scan to include the abdomen. Results showed most participants supported this addition, and the number of serious findings was similar to those detected in UK breast or bowel cancer screening programmes.

However, the abdominal scan was only offered on the day of the lung scan, giving little time for people to consider their decision. The process also added too much time to be practical for widespread implementation.

This new study will:

* Test whether mentioning the possible abdominal scan in the initial LCS invitation affects participation in LCS assessments.
* Test new processes to assess if the abdominal scan can be added to the lung scan with minimal extra time.
* Check if participants can be split between the lung scan only group and lung and abdominal scan group using an approach called 'cluster randomisation'. This will be important in case a bigger trial is needed.
* See whether the additional processes are acceptable

People aged 55-70 who are invited to the lung cancer screening will be eligible to take part in this study. Only those who are found to be at a high risk of lung cancer after their assessment, and therefore offered a lung scan, will be offered the abdominal scan, provided they have not had an abdominal scan in the previous 12 months or one booked in the next 3 months.

This study will take place in two existing lung cancer screening locations in Yorkshire.

ELIGIBILITY:
1. For the individual level randomisation to invitation control or invitation intervention

   Inclusion criteria: To be randomised at the individual level to receive an invitation letter for LCS (standard of care; invitation control) versus invitation letter for LCS with potential for an additional abdominal scan (invitation intervention):
   * Be eligible to be invited to the first round of a West Yorkshire and Harrogate LCS or a Humber and North Yorkshire Cancer Alliance LCS (i.e. have been identified as a smoker or ex-smoker and registered as living within the relevant LCS catchment area).
   * Be registered with a GP in England.
   * Be aged 55-70 years 364 days old at the date of invitation.

   Exclusion criteria

   • None
2. Eligibility criteria for the cluster level randomisation to scan intervention or scan control

   Inclusion criteria a): To be eligible for the cluster level randomisation the participant must:
   * Have been individually randomised to the invitation intervention arm
   * Have booked in for a LCS assessment

   Inclusion criteria b): To receive the CT Thorax plus ANCCT, the participant must:
   * Have been randomised to the scan intervention cluster
   * Be invited to attend for a LDCT Thorax based upon scores on either PLCOM2012 or Liverpool Lung Project (LLP) risk prediction models (PLCOM2012 risk of ≥1.51% over six years or LLPver2 five-year risk of ≥2.5%)14 during the LCS assessment.
   * Have attended the lung scan appointment
   * Have given electronic or written informed consent to participate

   Exclusion criteria

   Existing LCS exclusion criteria:
   * Participant does not have capacity to give consent (standard criteria for assessing capacity apply).
   * Weight or physical size exceeds restrictions for scanner (>200kg).
   * Participant unable to lie flat.
   * Poor physical fitness such that treatment with curative intent would be contra-indicated.
   * Participants who have had a full CT Thorax that meets the image reconstruction parameters of the programme in the last 12 months are not excluded from the lung screening programme, but would have their CT Thorax appointment deferred until 12 months have elapsed since that last scan, provided they still meet all inclusion criteria and have no exclusion criteria - if the deferred appointment is within the timeframe for TACTICAL1, they remain eligible but if deferred appointment is outside the timeframe for TACTICAL1 they would not be eligible.

   Additional TACTICAL1 exclusion criteria:

   • Had an abdominal CT in the previous 12 months or has one booked within the next 3 months.
   * For HNY, this is checked before the LCS assessment. Therefore, participants will be excluded before the LCS assessment.
   * For WYH, this is only checked after the LCS assessment. Therefore, anyone having had an abdominal CT in the previous 12 months or with one booked within the next 3 months will be excluded at this point (see 8.6).
3. Eligibility criteria for the process evaluation Health care professionals: Healthcare professionals involved in the delivery of LCS in any of the study areas who agree to take part.

Participants: People individually randomised to the invitation intervention arm who attend the LCS assessment or the scanning unit within the study period and who agree to be interviewed.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6272 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Attendance rate at the LCS phone call | 12 weeks after invitation letter is sent
  Attendance rate of the invitation intervention group to the LCS phone call is non-inferior to the attendance rate of the invitation control group and if so, whether it is superior.
Cluster randomisation assessment | At the point of LCS assessment, within 12 weeks of invitation
  Successful cluster randomisation of participants into scan control and scan intervention groups as demonstrated by groups of similar size.
Impact of abdominal scan on throughput | Up to 6 months after invitation
  Average number of participants scanned per standard LCS scanning day is no different when adding the ANCCT
Perceived impact of abdominal scan on throughput | Up to 6 months after invitation
  Data from daily short questionnaire completed by scanning unit staff shows perceived impact of TACTICAL activities on normal LCS processes is no different when ANCCT is added for at least 80% of days
Incremental time taken for each TACTICAL1 task compared with the existing LCS processes. | Up to 6 months after invitation
  The observed incremental time taken for each TACTICAL1 task compared with the existing LCS processes for a sub-sample of participants.
Over 75% of participants receiving abdominal scan are satisfied or very satisfied with their scanning unit experience | Up to 6 months after invitation
  Over 75% of participants are satisfied or very satisfied with their scanning unit experience as demonstrated by a post-scan feedback questionnaire.

SECONDARY OUTCOMES:
Percentage of participants taking up offer of abdominal scan | Up to 6 months after invitation.
  At least 80% of participants offered the ANCCT, accept the invitation and attend the scan

CONTACTS AND LOCATIONS:
Locations (1):
- Hull Teaching Hospitals Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No